CLINICAL TRIAL: NCT03054493
Title: Prevalence of Non-Nutritive Sucking Habits in a Group of Egyptian Children Aged 3-8 Years Old in Giza Governorate: A Cross Sectional Study.
Brief Title: Prevalence of NNSH in a Group of Egyptian Children Aged 3-8 Years Old in Giza Governorate: A Cross Sectional Study.
Acronym: NNSH
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Afnan Mohammad Nassar, Master dental student, pediatric dentistry department, Cairo University
Other Study IDs: AMNassar
Record Dates: First submitted 2017-02-11; First posted 2017-02-15 (Actual); Last update posted 2017-02-16 (Actual); Status verified 2017-02

CONDITIONS: Child Behavior
MeSH Terms: conditions — Child Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional

INTERVENTIONS:
Behavioral: no intervention — no intervention

SUMMARY:
1. Prevalence of non-nutritive sucking habits (NNSH) in a group of Egyptian children aged 3-8 years old in Giza Governorate.
2. Assessment of factors associated with NNSH.

DETAILED DESCRIPTION:
Several studies have reported on the prevalence of non-nutritive sucking behaviors among infants and young children in different populations. Non-nutritive sucking is regarded as a normal part of development, and early studies of its prevalence generally found that 70-90% of children had some history of a non-nutritive sucking habit. Like these early studies, most recent studies have used retrospective methods to assess the prevalence of non-nutritive sucking habits.

Prolonged duration of non-nutritive sucking behaviors may have consequences in regard to the developing orofacial structures and occlusion. Little is known as to why some children have sucking habits beyond the first 2 to 3 years of life.

Prevalence of NNSH and associated factors in Egyptian children might be different.

ELIGIBILITY:
Inclusion Criteria:

* 3-8 years old children.
* Children free of systemic diseases.
* Positive patient/parents acceptance for participation in the study.
* Both sexes will be included.

Exclusion Criteria:

* Disabled children.
* Children with cleft lip & palate.
* TMJ disorders.
* Children undergoing orthodontic/orthopedic treatment.
* Participants who were exposed to thumb sucking prevention programs.

Ages: 3 Years to 8 Years | Sex: All
Age Groups: Child
Study Population: A group of Egyptian children aged 3-8 years in Giza Governorate.
Sampling Method: Probability Sample
Enrollment: 1023 (Actual)
Dates: Start 2017-02-10 (Actual); Primary Completion 2017-06 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
non-nutritive sucking habits | 20 mins
  child sucking one or more of his/her digits and/or object beyond 36 months old.

CONTACTS AND LOCATIONS:
Overall Officials: Afnan Mo Nassar, Bechlor, Principal Investigator — Cairo University
Locations (1):
- Afnan Mohammad Nassar, 6th of October City, October 6, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Holanda AL, dos Santos SA, Fernandes de Sena M, Ferreira MA. Relationship between breast- and bottle-feeding and non-nutritive sucking habits. Oral Health Prev Dent. 2009;7(4):331-7. PMID 20011750
- [Background] Maia-Nader M, Silva de Araujo Figueiredo C, Pinheiro de Figueiredo F, Moura da Silva AA, Thomaz EB, Saraiva MC, Barbieri MA, Bettiol H. Factors associated with prolonged non-nutritive sucking habits in two cohorts of Brazilian children. BMC Public Health. 2014 Jul 22;14:743. doi: 10.1186/1471-2458-14-743. PMID 25053157
- [Background] Medeiros AP, Ferreira JT, Felicio CM. Correlation between feeding methods, non-nutritive sucking and orofacial behaviors. Pro Fono. 2009 Oct-Dec;21(4):315-9. doi: 10.1590/s0104-56872009000400009. PMID 20098950